CLINICAL TRIAL: NCT02405286
Title: Prospective Assessment of the Rockall Risk ScoringSystem in Patients With Upper Gastrointestinal Hemorrhage
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Iman Fawzy Montasser, Lecturer of tropical medicine , Ain Shams university, Ain Shams University
Other Study IDs: Rockall score
Record Dates: First submitted 2015-03-24; First posted 2015-04-01 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Gastrointestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Upeer gastrointestinal bleeding: * Adult Egyptian patients.
  * Patients with acute upper G.I hemorrhage.
  * Informed consent.
  Interventions: Other: Upper gastrointestinal endoscopy

INTERVENTIONS:
Other: Upper gastrointestinal endoscopy — Upper gastrointestinal endoscopy, if stigmata of recent hemorrhage are seen, varices are either injected with ethanolamine or banded, depending on the clinical setting and availability .

SUMMARY:
This study aimed to Assess the validity of the Rockall score for the prediction of rebleeding and death in patients with upper gastrointestinal bleeding.

DETAILED DESCRIPTION:
This present study aimed to evaluate:

Assess the validity of the Rockall score for the prediction of rebleeding and death in patients with upper gastrointestinal bleeding.

1- Technical Design: The technical design included research design, setting, subject and tools for data collection.

Research design:

A descriptive exploratory design was followed to achieve the aim of the study. Study setting: This study was conducted between Tropical department in AinShams university and Gastroenterology and Hepatology department in TheodorBilharz Research Institute.

Sample size: EPI - INFO program version 6 was used for sample size calculation guided by power of the test = 80% - confidence level =95% and accepted margin of error = 5% and risk ratio = 5.5 - total sample minimum accepted = 50 This study included 50 recipients and done Tropical department in Ain Shams university and Gastroenterology and Hepatology department in .

Theodore Bilharz Research Institute

ELIGIBILITY:
Inclusion Criteria:

* Adult Egyptian patients.
* Patients with acute upper G.I hemorrhage.
* Informed consent.

Exclusion Criteria:

* Refuse to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Egyptian patients with acute upper gastrointestinal bleeding
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Clinical condition of the patients with accute upper gastrointstinal bleeding after 48 hours from endoscopy | 48 hours

SECONDARY OUTCOMES:
number of participants with variceal bleeding and other causes of upper gastrointestinal bleeding regarding the clinical condition after 48 hours | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Egypt Ain Shams center University Hospitals, Cairo, Egypt